CLINICAL TRIAL: NCT01708187
Title: The Role of Cryopreserved Human Amniotic Membrane in the Surgical Repair of Peroneal Tendons: An Infrared Thermography Model
Brief Title: The Role of C-HAM in the Surgical Repair of Peroneal Tendons: An Infrared Thermography Model
Acronym: Amniox
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Protocol halted due to less than anticipated recruitment.
Sponsor: Orthopedic Foot and Ankle Center, Ohio (Other)
Responsible Party: Principal Investigator, Greg Berlet, MD, Orthopedic Foot and Ankle Center, Ohio
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OH1-12-00396
Record Dates: First submitted 2012-09-05; First posted 2012-10-16 (Estimated); Results first posted 2016-05-19 (Estimated); Last update posted 2016-11-03 (Estimated); Status verified 2016-09

CONDITIONS: Tendon Tears
Keywords: Peroneal tendon
MeSH Terms: interventions — Transplantation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Clarix™1k graft (Experimental): Group 1 will have standard peroneal repair surgery with the addition of the Clarix™1k tissue.
  Interventions: Biological: Clarix™1k graft
- Control arm without Clarix™1k graft (No Intervention): Group 2 will have standard peroneal repair surgery without the use of the Clarix™1k tissue.

INTERVENTIONS:
Biological: Clarix™1k graft — Group 1 will have standard peroneal repair surgery with the addition of the Clarix™1k tissue.
  Group 2 will have standard peroneal repair surgery without the use of the Clarix™1k tissue.
  Other Names: cryopreserved Human Amniotic Membrane (C-HAM) graft
  Arms: Clarix™1k graft

SUMMARY:
Peroneal tendon tears are a common etiology encountered by foot and ankle surgeons. Like all flexor tendon repairs adhesions are one of the more common challenges after surgery. Peroneal tendon gliding is key to their function as effective plantar flexors and evertors of the hindfoot. Scarring and adhesion correlate directly with the amount of inflammatory reaction at the wound site (Adzick 1994). Our goal is to have a surgical technique that allows for standard suture repair of the tendon yet allows for smooth gliding of the tendon with minimal adhesions. A prospective review on the surgical repair of the peroneal tendons utilizing Clarix™1k (Amniox Medical, Marietta, GA), cryopreserved Human Amniotic Membrane (C-HAM) graft will be performed. The investigators hypothesize that the use of cryopreserved Human Amniotic Membrane in conjunction with a peroneal tendon repair will decrease that amount of inflammation, overall recovery time of surgically repaired peroneal tendon tears, and adhesions.

ELIGIBILITY:
Inclusion Criteria:

1. Patients requiring surgical repair of the peroneal tendon
2. Patients who voluntarily consent to research participation
3. Patients over the age of 18

Exclusion Criteria:

1. Patients who display a high surgical risk as determined by the investigative surgeon
2. Previous surgical repair of the peroneal tendon less than 2 years prior to surgery
3. Peroneus brevis tears in zone 3 or 4 that may hinder recovery in the investigator's opinion
4. Patients with allergy or history of drug reactions to Ciprofloxacin or Amphotericin B
5. Patients who are pregnant or breast feeding.
6. Patients who have had a clinically diagnosed autoimmune disease
7. Patients who are unwilling to restrict pre and postoperative anti-inflammatories with the exception of ecotrin 325 mg QD for DVT prophylaxis during the postoperative immobilization period
8. Patients with an active infection
9. Patients who have a medical history that would likely make the patient an unreliable research participant
10. Patients requiring surgical repair of the peroneus longus tendon

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2012-10; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory C Berlet, MD, Principal Investigator — Orthopedic Foot and Ankle Center
Locations (1):
- Orthopedic Foot and Ankle Center, Westerville, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Clarix™1k Graft: Group 1 received standard peroneal repair surgery with the addition of the Clarix™1k tissue.
- Control Arm Without Clarix™1k Graft: Group 2 received standard peroneal repair surgery without the use of the Clarix™1k tissue.
Period: Overall Study
Arm/Group | Clarix™1k Graft | Control Arm Without Clarix™1k Graft
Started | 1 | 1
Completed | 1 | 0
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Clarix™1k Graft | Control Arm Without Clarix™1k Graft | Total
Number analyzed (Participants) | 1 | 1 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Ankle Pain, Inflammation, Function & Activity Limitation From Baseline to 12 Months
Description: Ankle pain measured via visual analog scale (VAS), function measured by American Orthopaedic Foot and Ankle Society (AOFAS) ankle hindfoot scale and Foot Function Index (FFI), activity limitation measured by AOFAS scale. Images taken via thermal camera to measure inflammation were not interpretable.
  VAS pain scale: 0-100, with a lower number representing a better score FFI scale: 0-100, with a lower number representing a better score AOFAS scale: 0-100, with a higher number representing a better score
Time Frame: Baseline,12 months
Measure: Number; unit: units on a scale
Arm/Group | Clarix™1k Graft | Control Arm Without Clarix™1k Graft
Number analyzed (Participants) | 1 | 0
units on a scale
  VAS pain at Baseline | 66 |
  VAS pain at 12 months | 0 |
  Change in VAS pain from Baseline to 12 months | -66 |
  FFI at Baseline | 61.76 |
  FFI at 12 months | 4.71 |
  Change in FFI from Baseline to 12 months | -57.05 |
  AOFAS at Baseline | 70 |
  AOFAS at 12 months | 90 |
  Change in AOFAS from Baseline to 12 months | 20 |

ADVERSE EVENTS:
Arm/Group | Clarix™1k Graft | Control Arm Without Clarix™1k Graft
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 1/1 | 0/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clarix™1k Graft (N=1) | Control Arm Without Clarix™1k Graft (N=1)
Herpes Zoster (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Early termination leading to only one subject completing the trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No